CLINICAL TRIAL: NCT06542913
Title: Left Lobe Versus Right Lobe in Adult Living Donor Liver Transplantation in Borderline GRWR: Prospective Cohort Study
Brief Title: Left Lobe Versus Right Lobe in Adult Living Donor Liver Transplantation in Borderline GRWR
Acronym: LDLT
Status: Not yet recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: ltvsrtldlt; Ain Shams University (Other: Ain Shams University)
Record Dates: First submitted 2024-08-03; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Liver Transplant; Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- right lobe: cases underwent LDLT for right lobe with borderline GRWR
- left lobe: cases underwent LDLT for left lobe with borderline GRWR

SUMMARY:
a prospective cohort study comparing outcomes of left lobe and right lobe adult living donor liver transplantation

ELIGIBILITY:
Inclusion Criteria:

* GRWR below 1

Exclusion Criteria:

* patients with renal impairment portal vein thrombosis vascular complications

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients presented to our center for LDLT
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
small for size syndrome | 1 year
  small for size syndrome

SECONDARY OUTCOMES:
other complications after LDLT | 1 year
  other complications after LDLT

IPD SHARING:
Plan to Share IPD: Undecided